CLINICAL TRIAL: NCT01157013
Title: The Role of Positron Emission Tomography (PET) Imaging in the Evaluation of Response to Sorafenib Treatment in Advanced Hepatocellular Carcinoma.
Brief Title: Role of Positron Emission Tomography in the Evaluation of Response to Sorafenib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Carlos III Health Institute (Other Government); Spanish National Health System (Other); Aragon Health Science Institute (Other Government)
Responsible Party: Roberto A. Pazo Cid, MD, Aragon Health Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI09/90721; ETES08/90721 (Other Grant/Funding Number: ETES 09/9072 Fondo de Investigaciones Sanitarias, Spain)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Positron Emission Tomography; Hepatocellular carcinoma; Liver Cancer; Sorafenib; Response Evaluation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced Hepatocellular Carcinoma (Experimental): Hepatocellular carcinoma patients not candidates to local and/or curative treatment and an expected overall survival of at least three months and who are susceptible of receiving sorafenib therapy.
  Interventions: Other: Positron emission tomography with fludeoxyglucose F 18

INTERVENTIONS:
Other: Positron emission tomography with fludeoxyglucose F 18 — Patients receive fludeoxyglucose F 18 (^18FDG) IV. Beginning 1 hour later, patients undergo whole-body positron emission tomography (PET) scanning. Patients also undergo conventional radiographic staging of their disease.
  Other Names: PET

SUMMARY:
Positron emission tomography (PET) with [18F]fluorodeoxyglucose (FDG-PET) evaluates cancer cell glycolysis(Warburg effect) as a surrogate for tumor response.The hypothesis of this study is that early changes in FDG-PET signal can predict sorafenib response in hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a major health issue worldwide, particularly in Asia and Africa, and a disease that has increased in incidence in the Western world over the past 20 years primarily as a result of the prevalence of hepatitis C virus infection, which predisposes patients to HCC.

Sorafenib (a new oral potent multikinase inhibitor directed against both tumour proliferation and angiogenesis) can be considered standard of care for patients with advanced and metastatic HCC who are not candidates for curative or locoregional therapies. Clinical benefit has been shown in 75% of patients with advanced HCC.

PET is a noninvasive imaging technique which might be an effective tool for evaluating sorafenib treatment in HCC. The aim of this study is to evaluate this new treatment with PET with fluorodeoxyglucose (FDG), since the use of only computed tomography (CT) measurements can be questioned. Our hypothesis is that early effects of sorafenib treatment in advanced HCC can be detected and quantified by PET-CT after one month of treatment. We try to reveal a decrease in tumour glucose uptake at one month and correlate it with other radiologic findings (measured by CT and diffusion-weighted nuclear resonance imaging) and the more clinically relevant endpoints clinical benefit and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* advanced hepatocellular carcinoma: diagnostic assessment by biopsy/cytology; in cirrhotic patients conventional radiologic criteria are also accepted
* more than 18 years of age.
* life expectancy greater than three months
* candidate to sorafenib therapy
* informed consent required

Exclusion Criteria:

* hepatocellular carcinoma patients candidate to local/curative therapies(surgery/radiofrequency/TACE/other local therapy
* another active cancer than primary liver cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Response to sorafenib therapy shown in PET Scans | Baseline and after three weeks on treatment
  Changes in the SUVmax during treatment (SUVmax) were determined by the following equation: (post-treatment SUVmax - baseline SUVmax)/baseline SUVmax, expressed in percentage. The SUVmax for all target lesions were averaged(mSUVmax) and reported per the 1999 European Organisation for Research and Treatment of Cancer recommendations.

SECONDARY OUTCOMES:
Tumor response evaluated by CT and MRI | Basal and every two months
  Tumor response was reported per Response Evaluation Criteria in Solid Tumors (RECIST) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Roberto A. Pazo Cid, MD, Principal Investigator — Aragon Health Institute. Hospital Miguel Servet
Locations (1):
- Miguel Servet University Hospital, Zaragoza, Aragon, Spain

REFERENCES:
- See also: Red Tematica de Investigacion Cooperativa en Cancer. Hospital Universitario Miguel Servet — http://www.rticcc.org/articulos/quienessomos/nodos/mservet.shtml